CLINICAL TRIAL: NCT07000084
Title: GAIN-BCG: Gemcitabine Alternating With INtravesical BCG Randomized Against BCG Alone for Patients With Recurrent High Grade Non-Muscle Invasive Bladder Cancer
Brief Title: Testing the Addition of an Anti-Cancer Drug, Gemcitabine, to Usual Treatment (BCG Alone) in People Whose Non-Muscle Invasive Bladder Cancer (NMIBC) Came Back After Prior BCG Therapy
Acronym: GAIN-BCG
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A032303; NCI-2025-02655 (Registry Identifier: NCI Clinical Trial Reporting Program)
Record Dates: First submitted 2025-05-23; First posted 2025-05-31 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Recurrent Non-Muscle Invasive Bladder Carcinoma; Stage 0a Bladder Cancer AJCC v8; Stage I Bladder Cancer AJCC v8
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms | interventions — Cystoscopy; Magnetic Resonance Spectroscopy; Transurethral Resection of Bladder; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (BCG) (Active Comparator): Patients receive BCG intravesically over 2 hours QW for 6 weeks. 2-6 weeks after completing endoscopic assessment, patients receive BCG over 2 hours QW for 3 weeks at month 3, 6 and 12 in the absence of disease progression or unacceptable toxicity. Patients undergo bladder biopsy, TURBT, cystoscopy, CT scan/MRI and blood and urine sample collection throughout the study.
  Interventions: Biological: BCG Solution; Procedure: Biopsy of Bladder; Procedure: Cystoscopy; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Biospecimen Collection; Procedure: Transurethral Resection of Bladder Tumor
- Arm B (BCG and gemcitabine) (Experimental): Patients receive gemcitabe intravesically over 1 hour twice weekly on weeks 1 and 10 and once weekly on weeks 4 and 7. Patients also receive BCG intravesically over 2 hours QW on weeks 2, 3, 6, 8 and 9. 2-6 weeks after completing endoscopic assessment, patients receive gemcitable intravesically over 1 hour on week 1 and BCG intravesically over 2 hours on week 2-4 at month 3, 6 and 12 in the absence of disease progression or unacceptable toxicity. Patients undergo bladder biopsy, TURBT, cystoscopy, CT scan/MRI and blood and urine sample collection throughout the study.
  Interventions: Biological: BCG Solution; Procedure: Biopsy of Bladder; Procedure: Cystoscopy; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Biospecimen Collection; Procedure: Transurethral Resection of Bladder Tumor; Drug: Gemcitabine

INTERVENTIONS:
Biological: BCG Solution — Given intravesically
  Other Names: Bacillus Calmette Guerin Solution
Procedure: Biopsy of Bladder — Undergo bladder biopsy
  Other Names: Bladder Biopsy
Procedure: Cystoscopy — Undergo cystoscopy
Procedure: Computed Tomography — Undergo CT Scan
  Other Names: CAT Scan; CT Scan
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: MRI
Procedure: Biospecimen Collection — Undergo blood and urine sample collection
Procedure: Transurethral Resection of Bladder Tumor — Undergo TURBT
  Other Names: TURBT
Drug: Gemcitabine — Given intravesically
  Arms: Arm B (BCG and gemcitabine)

SUMMARY:
This phase III trial compares the effect of adding gemcitabine to intravesical Bacillus Calmette Guerin (BCG) versus intravesical BCG alone in patients with non-muscle invasive bladder cancer that has come back after a period of improvement (recurrent). Gemcitabine is a chemotherapy drug that blocks the cells from making deoxyribonucleic acid (DNA) and may kill cancer cells. Intravesical BCG is a solution containing the live BCG bacteria that is placed in the bladder via a catheter (intravesical). When the solution comes into direct contact with the bladder wall, it stimulates the body's immune system which kills tumor cells. Giving gemcitabine with intravesical BCG may kill more tumor cells in patients with recurrent non-muscle invasive bladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare high-grade recurrence-free-survival between treated with gemcitabine with BCG (GemBCG) compared to those treated with BCG alone.

SECONDARY OBJECTIVES:

I. To compare the proportion of patients who remain high grade cancer free on initial post-treatment cystoscopic biopsies/transurethral resection of bladder tumor (TURBT) (week 13/month 3) between those treated with GemBCG compared to those treated with BCG alone.

II. To compare the 6-month (Week 25) complete response rate and the complete response durability between patients treated with GemBCG compared to those treated with BCG alone among patients with pre-treatment CIS.

III. To compare the time to recurrence of any-grade bladder cancer between patients treated with GemBCG compared those treated with BCG alone.

IV. To compare the progression-free-survival between patients treated with GemBCG compared to those treated with BCG alone.

V. To compare the cystectomy-free-survival between patients treated with GemBCG compared to those treated with BCG alone.

VI. To compare the proportion of patients free from BCG-unresponsive NMIBC between those treated with GemBCG compared to those treated with BCG alone.

VII. To determine the safety of and toxicity associated with GemBCG treatment relative to that of BCG treatment alone.

EXPLORATORY OBJECTIVE:

I. To collect tumor tissue/bladder biopsies, blood, and urine samples for biobanking that will enable future correlative studies.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive BCG intravesically over 2 hours once per week (QW) for 6 weeks. 2-6 weeks after completing endoscopic assessment, patients receive BCG over 2 hours QW for 3 weeks at month 3, 6 and 12 in the absence of disease progression or unacceptable toxicity. Patients undergo bladder biopsy, TURBT, cystoscopy, computed tomography (CT) scan/ magnetic resonance imaging (MRI) and blood and urine sample collection throughout the study.

ARM B: Patients receive gemcitabe intravesically over 1 hour twice weekly on weeks 1 and 10 and once weekly on weeks 4 and 7. Patients also receive BCG intravesically over 2 hours QW on weeks 2, 3, 6, 8 and 9. 2-6 weeks after completing endoscopic assessment, patients receive gemcitable intravesically over 1 hour on week 1 and BCG intravesically over 2 hours on week 2-4 at month 3, 6 and 12 in the absence of disease progression or unacceptable toxicity. Patients undergo bladder biopsy, TURBT, cystoscopy, CT scan/MRI and blood and urine sample collection throughout the study.

After completion of study treatment, patients are followed every 3 months for 2 years, then every 6 months for 3 years up to 5 years from randomization.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of Disease: Histologic confirmation of urothelial carcinoma that is high grade Ta, high grade T1, or Tis (Tis/carcinoma in situ [CIS] only disease) within 120 days prior to randomization
* Any component of neuroendocrine carcinoma (i.e., small cell or large cell) is not allowed. Other histologic subtypes/variant histologies are allowed so long as there is a predominantly urothelial component.

  * Note: Pure squamous cell carcinoma or pure adenocarcinoma without a urothelial component are not allowed
* All visible papillary lesions must be macroscopically resected by TURBT within 90 days of randomization. (Residual CIS is permitted).

  * If the treating urologist did not perform the TURBT, the treating urologist must perform a cystoscopy within 45 days prior to randomization to confirm the absence of visible papillary disease
* All patients with high grade T1 must undergo a restaging TURBT within 90 days of randomization. Patients who undergo a restaging TURBT that shows no residual cancer in the specimen are still eligible for trial based on prior TURBT
* Patients must have BCG-Exposed non muscle invasive bladder carcinoma (NMIBC), defined as recurrent high grade NMIBC within 24 months of last BCG exposure but not meeting the definition of BCG unresponsive disease

  * Note: Up to 26 months from the last BCG instillation is allowed for the treating physician to perform a transurethral resection of bladder tumor (TURBT) so long as there is evidence/suspicion of recurrent disease (by positive cytology, imaging, or cystoscopy) within 24 months of last exposure to BCG.
  * Note: A patient who previously met the definition of BCG unresponsive NMIBC but no longer currently meets unresponsive criteria may still enroll in this trial so long as the treating urologist believes re-treatment with BCG is a reasonable treatment option for that patient.
  * BCG-exposed NMIBC criteria is defined as:

    * Any high grade NMIBC recurrence within 24 months of induction only BCG, or
    * A high grade papillary NMIBC (Ta/T1) recurrence between 6-24 months of last exposure to induction + maintenance BCG, or
    * A high-grade CIS (with or without Ta/T1 papillary disease) recurrence within 12-24 months of last exposure to induction + maintenance BCG.
  * Patient must not have BCG-unresponsive NMIBC, defined as:

    * Persistent or recurrent high-grade papillary NMIBC (Ta/T1) < 6 months of "adequate" BCG, or
    * A high-grade CIS (with or without Ta/T1 papillary disease) recurrence < 12 months of "adequate" BCG, or
    * A high grade T1 recurrence at the first 3-month assessment from induction BCG
    * "Adequate" BCG is defined as ≥5 of 6 doses of induction BCG therapy with either

      * ≥ 2 of 3 doses of maintenance BCG, or
      * ≥ 2 of planned 6 instillations of repeat induction BCG given within a 6 month time period
* More than one prior induction course of BCG and/or prior maintenance BCG is allowed so long as the patient does not currently met the definition of BCG unresponsive disease
* Prior treatment with any intravesical chemotherapy (both perioperative and induction course) for NMIBC is allowed, including gemcitabine either alone or in combination (ie. gemcitabine plus docetaxel) or gemcitabine delivered through a intravesical delivery system (ie. TAR-200)
* Prior treatment with any systemic or intravesical agents for NMIBC is allowed, regardless of whether it is given either alone or in prior combination with BCG (ie. Prior treatment with pembrolizumab, other immune checkpoint inhibitors, nadofaragene firadenovec, nogapendekin alfa inbakicept, cretostimogene grenadenorepvec, etc. are all allowed)
* Patients must not have a history of intolerance to BCG (ie needing to stop BCG induction or maintenance due to toxicity) or intolerance to any other intravesical therapies
* Patients must not have compromised bladder function such that they are unlikely to tolerate further intravesical therapies
* Patient must not have any prior history or current evidence of muscle-invasive (i.e., T2, T3, T4), locally advanced unresectable, or metastatic urothelial carcinoma as assessed on radiographic imaging obtained within 120 days prior to randomization.

  * The radiographic imaging includes a CT Scan or MRI of the abdomen/pelvis with intravenous contrast, with a CT or MRI urogram preferred. If a patient is unable to receive intravenous contrast due to renal function or allergy, then either a CT scan or MRI of the abdomen/pelvis without intravenous contrast is acceptable
* Patients with a history of upper tract urothelial carcinoma are allowed so long as they had localized non-muscle invasive (Ta, T1, Tis) that has been definitively treated with surgery (nephroureterectomy or ureterectomy) with at least one post-treatment disease assessment imaging study that demonstrates no evidence of residual upper tract disease
* Patients with a history of, or current evidence of, non-invasive (Ta/Tis) urothelial carcinoma of the prostatic urethra are eligible so long as a transurethral resection of prostate (TURP) is performed before enrollment and there is prostatic glandular tissue without evidence of lamina propria invasion or prostatic stromal invasion
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* Age ≥ 18 years
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Not pregnant and not nursing, Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used. All patients of childbearing potential must have a blood test or urine study within 14 days prior to randomization to rule out pregnancy. A patient of childbearing potential is defined as anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria:

  * has achieved menarche at some point
  * has not undergone a hysterectomy or bilateral oophorectomy
  * has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2028-06-05 (Estimated); Study Completion 2028-12-05 (Estimated)

PRIMARY OUTCOMES:
High Grade Recurrence-free survival (HG-RFS) | Up to 5 years
  HG-RFS will be calculated from randomization until the detection of a high-grade bladder cancer recurrence (biopsy proven intravesical recurrence or distant metastasis), cystectomy, or death, whichever occurs first. Patients who are alive and without documented high-grade recurrence will be censored at the time of last disease evaluation. HG-RFS will be compared between the two study arms using a stratified log-rank test. The treatment effect will be estimated with a hazard ratio (HR) and corresponding 95% confidence interval obtained from a stratified Cox model with treatment group (

SECONDARY OUTCOMES:
High-grade cancer free at 3 months | at 3 months
  A patient will be classified as being cancer free if no high-grade bladder cancer is detected upon a cystoscopic biopsy (± transurethral resection of bladder tumor [TURBT]). This will be calculated as the number of patients who underwent cystoscopic biopsy with or without TURBT at 3 months and no high-grade cancer was detected, divided by the total number of patients.
6-month Complete Response | At 6 months
  Complete response rate will be determined among patients who had carcinoma in situ (CIS) at baseline. Patients will be classified as having a complete response at 6 months if there is no biopsy-proven high grade bladder cancer detected based on a cystoscopy and urinary cytology (± biopsy/TURBT). This will be calculated as the number of patients who had CIS at baseline and who had no evidence of disease at 6-months, divided by the total number of patients who had CIS at baseline. The proportion of patients who remain with a complete response will be compared between the two arms with a chi-square test or Fisher's exact test.
Durability of Response | Up to 5 years
  o Durability of the response will be determined only in the patients who had CIS at baseline and had a complete response at 6 months. This will be measured as time from the 6-month evaluation until documented disease recurrence, censoring patients without disease recurrence at time of death or at last disease evaluation, whichever is last. The durability of response will be compared between the two treatment groups using a log-rank test, and Kaplan-Meier estimators will be used to determine the median durability.
Recurrence-free survival | Up to 5 years
  Recurrence-free survival will be calculated as the time from randomization until the detection of any grade bladder cancer, censoring those without documented disease recurrence at time of last disease evaluation or death, whichever occurs last. This will be compared between the two treatment arms using a stratified log-rank test. An estimate of the outcome differences between the arms will be made with a HR and 95% confidence interval generated by a stratified Cox model.
Progression-free survival | up to 5 years
  Progression-free survival will be calculated as the time from randomization until disease progression, defined as development of muscle invasive disease (stage greater than or equal to T2), lymph node or distant metastasis, or death without documented disease progression. This will be compared between the two treatment arms using a stratified log-rank test. An estimate of the outcome differences between the arms will be made with a HR and 95% confidence interval generated by a stratified Cox model.
Cystectomy-free survival | up to 5 years
  Cystectomy-free survival will be defined as the time from randomization until the patient undergoes a cystectomy, censoring patients without a cystectomy at last follow-up or death, whichever is last. This will be compared between the two treatment arms using a stratified log-rank test. An estimate of the outcome differences between the arms will be made with a HR and 95% confidence generated by a stratified Cox model.
• Bacille Calmette Guerin (BCG)-unresponsive non muscle invasive bladder cancer free survival | up to 5 years
  BCG unresponsive NMIBC free survival will be defined as time from randomization until the patient develops BCG unresponsive NMIBC, defined as persistent or recurrent high-grade papillary NMIBC (Ta/T1) <6 months of "adequate" BCG (≥5 of 6 plus an additional ≥2 doses of BCG) or CIS (with or without Ta/T1 papillary disease) recurrence <12 months of "adequate" BCG (≥5 of 6 plus an additional ≥2 doses of BCG) or High Grade T1 at week 13 (month 3) assessment. Patients who do not develop BCG-unresponsive NMIBC will be censored at the time of their last follow-up or death, whichever is last. This will be compared between the two treatment arms using a stratified log-rank test. An estimate of the outcome differences between the arms will be made with a HR and 95% confidence interval generated by a stratified Cox model.
Rate of Grade 3+ Adverse Events | Up to 5 years
  o Adverse events will be collected and graded according to the NCI Common Terminology Criteria for Adverse Events version 5.0. The number (percent) of patients that experience each grade 3+ adverse event will be summarized by treatment arm. In addition, the number (percent) of patients that experience a grade 3+, grade 4+, and grade 5 adverse event will be summarized by treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Pietzak, MD, Study Chair — Alliance for Clinical Trials in Oncology
Locations (53):
- United States (53):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Marjorie Weinberg Cancer Center at Loyola-Gottlieb, Melrose Park, Illinois
  - IU Health West Hospital, Avon, Indiana
  - IU Health North Hospital, Carmel, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Mary Bird Perkins Cancer Center - Metairie, Metairie, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - FMH James M Stockman Cancer Institute, Frederick, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Hi-Line Sletten Cancer Center, Havre, Montana
  - Benefis Helena Specialty Center, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Cancer Center Dickson City, Dickson City, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center-Rockledge, Rockledge, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Memorial Hospital of Laramie County, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming